CLINICAL TRIAL: NCT02648399
Title: Prospective Study on the Clinical Prognosis of Bilateral Central Lymph Node Dissection in the Patients With Unilateral Thyroid Papillary Carcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, wenxin zhao, Director,Vise Head of Acscular and Thyroid Department,Principal Investigator, Clinical Professor, Fujian Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: wzhao
Record Dates: First submitted 2015-12-13; First posted 2016-01-07 (Estimated); Last update posted 2016-01-07 (Estimated); Status verified 2016-01

CONDITIONS: Thyroid Papillary Carcinoma
Keywords: thyroid carcinoma; center lymph node dissection
MeSH Terms: conditions — Thyroid Cancer, Papillary; Thyroid Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- control group (Placebo Comparator): only unilateral center lymph node dissection
  Interventions: Procedure: surgery：UCND（unilateral central lymph node dissection）
- experimental group (Experimental): bilateral center lymph node dissection
  Interventions: Procedure: surgery：BCND（bilateral central lymph node dissection）

INTERVENTIONS:
Procedure: surgery：BCND（bilateral central lymph node dissection）
  Other Names: aad another central lymph node dissection
  Arms: experimental group
Procedure: surgery：UCND（unilateral central lymph node dissection）
  Other Names: only unilateral central lymph node dissection
  Arms: control group

SUMMARY:
This study recruit the patients with unilateral papillary thyroid cancer before operation,the patients agree to enter the test,and divided into experimental and control group.experimental group patients receive the surgery including unilateral thyroid lobectomy and bilateral central lymph node dissection.and control group receive the surgery including unilateral thyroid lobectomy and unilateral central lymph node dissection.last the investigators compare numbers of patient with tumor recurrence and metastasis rate of 5 years,numbers of metastatic lymph node,and numbers of participants with adverse events related to treatment between two groups in order to evaluate the significance of bilateral lymph node dissection.

ELIGIBILITY:
according by thyroid carcinoma TNM(tumor,lymph node, metastasis) staging of NCCN (National Comprehensive Cancer Network)

Inclusion Criteria:

* 1.Unilateral thyroid papillary carcinoma 2.TNM staging: T1~2N0M0

Exclusion Criteria:

* 1.Bilateral thyroid papillary carcinoma 2.isthmus thyroid carcinoma 3.TNM staging: T3orT4 4.Clinic N1orM1

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 300 (Estimated)
Dates: Start 2015-12; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
tumor recurrence | 5 years
  numbers of patients with tumor recurrence
numbers of metastatic lymph node | 1 years
  numbers of metastatic lymph node
adverse events related to treatment | 1 years
  numbers of participants with adverse events including recurrent nerve injury，parathyroid injury，hemorrhage

SECONDARY OUTCOMES:
relations between the lymph metastasis and TNM staging | 1 years
  Coefficient R (SPSS software for correlation analysis)
relations between the lymph metastasis and tumor location | 1 years
  Coefficient R (SPSS software for correlation analysis)

CONTACTS AND LOCATIONS:
Overall Officials: wenxin zhao, doctor, Principal Investigator — Fujian Medical University Union Hospital
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No